CLINICAL TRIAL: NCT00976781
Title: Identifying the Gaps in the Diagnosis and Management of Hepatitis C
Status: Withdrawn | Type: Observational
Why Stopped: Decision not to move forward. Lack of funding.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: IRB no. 4775
Record Dates: First submitted 2009-09-10; First posted 2009-09-14 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify the gaps in diagnosing and managing hepatitis C infected patients so that interventions can be targeted to address these problem areas in order to optimize care of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Every patient diagnosed with hepatitis C

Exclusion Criteria:

* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
This is a retrospective observational study. The outcome measure would be the number of patients who are actually followed and treated for hepatitis C after they have been diagnosed | One year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Hnery Ford Hospital, Detroit, Michigan